CLINICAL TRIAL: NCT05196360
Title: A Phase I Study to Evaluate the Safety, Tolerability and Pharmacokinetic Characteristics of MAX-10181 in Patients With Advanced Solid Tumor
Brief Title: MAX-10181 in Patients With Advanced Solid Tumor
Acronym: PD-L1
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Maxinovel Pty., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MAX-10181-002; MAX-10181 (Other: Maxinovel)
Record Dates: First submitted 2021-10-13; First posted 2022-01-19 (Actual); Last update posted 2022-01-19 (Actual); Status verified 2022-01

CONDITIONS: Solid Tumor
Keywords: PD-1/L1; immunotherapy; advanced solid tumors

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- MAX-10181 (Experimental): tables
  Interventions: Drug: MAX-10181

INTERVENTIONS:
Drug: MAX-10181 — Part 1: Dose escalation, MAX-10181 once or twice daily with dose modifications based on tolerability criteria.
  Part 2: Dose expansion, Recommended doses from Part 1.

SUMMARY:
This is a multi-center, open-label, single-arm, dose-escalation Phase I study to evaluate the safety and tolerability of MAX-10181 in patients with advanced solid tumor.

DETAILED DESCRIPTION:
This is a multi-center, first-in-human, non-randomized, open-label, single-arm, dose-escalation Phase I study to evaluate the safety and tolerability of MAX-10181 in patients with advanced solid tumors.

ELIGIBILITY:
Inclusion Criteria:

* Males and/or females over age 18.
* Histologically or cytologically confirmed advanced or metastatic solid tumor for -which no established standard therapy is available.
* At least one measurable lesion by CT or MRI according to RECIST1.1, which is not in irradiated area (only for expansion phase).
* Recovered from toxicities of prior anti-cancer treatment to Grade 1 or less (in case of alopecia, Grade 2 is acceptable).
* Life expectancy of at least 3 months.
* Female participants of child bearing potential agree not to be pregnant or lactating during the study and for three months following the last dose of study drug. Both men and women of reproductive potential must agree to use a highly effective method of birth control during the study and for three months following the last dose of study drug. A highly effective method of contraception is defined as one that results in a low failure rate, i.e., less than 1% per year, when used consistently and correctly.

Exclusion Criteria:

* Laboratory values not within the Protocol-defined range.
* Cardiac disease with New York Heart Association (NYHA) Class III or IV, including congestive heart failure, myocardial infarction within 6 months prior to the trial entry, unstable arrhythmia, or symptomatic peripheral arterial vascular disease.
* Previously treated malignancies other than the current disease, except for adequately treated non-melanoma skin cancer, in situ cancer, or other cancer from which the subject has been disease-free for at least 5 years at the trial entry.
* Active, uncontrolled bacterial, viral, or fungal infections, requiring systemic therapy.

Major surgery, other than diagnostic surgery, within 4 weeks prior to the trial entry, without complete recovery.

* Medical history of difficulty swallowing, malabsorption or other chronic gastrointestinal disease, or conditions that may hamper compliance and/or absorption of the tested product.
* Anti-cancer treatment with radiation therapy, surgery, chemotherapy, targeted therapies (erlotinib, lapatinib, etc.), hormone therapy, or immunotherapy within 4 weeks (6 weeks for nitrosoureas or Mitomycin C) prior to trial entry.
* Known infection with human immunodeficiency virus (HIV), hepatitis B, or hepatitis C.
* History of upper gastrointestinal hemorrhage, peptic ulcer disease, or bleeding diathesis.
* History of organ allograft, autologous stem cell transplantation, or allogeneic stem cell transplantation.
* Concomitant disease or condition that could interfere with the conduct of the trial, or that would, in the opinion of the Investigator, pose an unacceptable risk to the subject in this trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2021-08-11 (Actual); Primary Completion 2023-01-01 (Estimated); Study Completion 2023-05-01 (Estimated)

PRIMARY OUTCOMES:
Adverse events (AEs) | 3 years
  Incidence of treatment-related AEs
Maximum tolerated dose (MTD） | 4 weeks
  MTD will be defined as the maximum dose level at which no more than 1 of 3 participants experience a dose-limiting toxicity (DLT) within the first 4 weeks of multiple dosing.
Phase II dose (RP2D) | 4 weeks
  The number and proportion of patients experiencing at least 1 dose-limiting toxicity (DLT) will be used as the primary measure to evaluate the RP2D of MAX-10181.

SECONDARY OUTCOMES:
Tmax | Approximately 4 weeks
  Time to maximum plasma concentration
Cmax | Approximately 4 weeks
  Time to maximum plasma concentration
  [Time Frame: Approximately 4 weeks]
AUC | Approximately 4 weeks
  Area under the time-concentration curve
t1/2 | Approximately 4 weeks
  Observed terminal half-life
Objective response rate (ORR) | 12 months (anticipated)
  The ORR is defined as the proportion of subjects with confirmed CR or confirmed PR, based on RECIST Version 1.1.

CONTACTS AND LOCATIONS:
Overall Officials: Yonghong Zhu, MD,Ph.D, Study Director — Maxinovel Pty., Ltd.
Locations (1):
- The First Affiliated Hospital, Zhejiang University, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: No